CLINICAL TRIAL: NCT06795971
Title: Effects of Face Mask Continuous Positive Airway Pressure Vs. Noninvasive Ventilation Vs. High-flow Nasal Oxygen on Intubation-free Survival in Acute Hypoxemic Respiratory Failure: the TRIPOD Randomized Clinical Trial
Acronym: TRIPOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIPOD Study
Record Dates: First submitted 2025-01-11; First posted 2025-01-28 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Acute Hypoxemic Respiratory Failure; High-Flow Nasal Oxygen Therapy; Noninvasive Ventilation; Continuous Positive Airway Pressure (CPAP)
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Continuous Positive Airway Pressure; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Continuous Positive Airway Pressure (Experimental): Patients will receive continuous positive airway pressure
  Interventions: Device: Continuous Positive Airway Pressure
- High-flow nasal oxygen (Active Comparator): Patients will receive high-flow nasal oxygen
  Interventions: Device: High-flow nasal oxygen
- Non-invasive ventilation (Active Comparator): Patients will receive non-invasive ventilation
  Interventions: Device: Non-invasive ventilation

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — 1. Patients were placed at a 45-degree supine position, and noninvasive ventilation was delivered to the patient through a face mask connected to an ICU ventilator.
  2. PEEP was started at 5 cm H2O with a FiO2 of 0.5 at initiation. PEEP and FiO2 were titrated to maintain SpO2 between 94 and 98%, remaining constant for at least 5 min.
  3. CPAP was initiated with a first session of at least 4 h, the minimally required duration of noninvasive ventilation was 16 hours per day for at least 2 calendar days. Between noninvasive-ventilation sessions, patients received HFNO.
  Arms: Continuous Positive Airway Pressure
Device: High-flow nasal oxygen — 1. Oxygen was passed through a heated humidifier (MR850, Fisher and Paykel Healthcare) and applied continuously through large-bore binasal prongs, with a gas flow rate of 50 liters per minute and an FiO2 of 0.5 at initiation. HFNO heating temperature was prespecified at 37°C.
  2. FiO2 will be titrated to maintain SpO2 between 94 and 98%, remaining constant for at least 5 min.
  3. HFNO was applied for at least 2 calendar days.
  Arms: High-flow nasal oxygen
Device: Non-invasive ventilation — 1. Patients were placed at a 45-degree supine position, and noninvasive ventilation was also delivered to the patient through a face mask connected to an ICU ventilator. The mask most appropriate for the patient will be selected and adjusted to minimize leakage and pressure points.
  2. The inspiratory positive airway pressure (pressure support plus PEEP) was initiated between 12 and 14 cm H2O, PEEP was started at 5 cm H2O with a FiO2 of 0.5 at initiation. FiO2 was titrated to maintain SpO2 between 94 and 98%, remaining constant for at least 5 min.
  3. NIV was initiated with a first session of at least 4 h, the minimally required duration of noninvasive ventilation was 16 hours per day for at least 2 calendar days. Between noninvasive-ventilation sessions, patients received HFNO.
  Arms: Non-invasive ventilation

SUMMARY:
Acute hypoxemic respiratory failure (AHRF) is a common indication for admission to an intensive care unit (ICU), with mortality exceeding 50% in cases where invasive mechanical ventilation is needed. Therefore, assessment of the most adequate oxygen strategy to avoid intubation in patients with AHRF deserves consideration.Previous studies have indicated that non-invasive oxygenation strategies, including high-flow nasal oxygen (HFNO), helmet or face mask noninvasive ventilation (NIV), and continuous positive airway pressure (CPAP), are effective in preventing endotracheal intubation in adult patients with AHRF when compared to the standard oxygen therapy. However, the optimal non-invasive oxygenation strategies remain uncertain. This study aim to determine whether CPAP, compared with HFNC or NIV, increase the intubation-free survival during study period in patients with AHRF.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 yrs;
2. A ratio of the partial pressure of arterial oxygen (PaO2) to the FiO2 of 300 mm Hg or less, or a ratio of pulse oximetry oxygen saturation (SpO2) to the FiO2 of 315 or less (SpO2≤97%) and the need for (1) noninvasive positive pressure ventilation with at least 5 cm H2O PEEP, or (2) high-flow nasal cannula at 30L/min or higher, or (3) standard oxygen with oxygen flow rate of at least 10 L/min;
3. Sign informed consent.

Exclusion Criteria:

1. Patients that have already received Continuous positive airway pressure, Noninvasive ventilation continuously for more than 24 hours before the screening visit.
2. Previous bout of mechanical ventilation during index hospitalization.
3. Exacerbation of chronic lung disease, including asthma or chronic obstructive pulmonary disease.
4. Moderate to severe cardiac insufficiency (New York Heart Association class >II or left ventricular ejection fraction<50%) or cardiogenic pulmonary edema.
5. Hemodynamic dysfunction, defined as vasopressor dose > 0.3 µg/kg/min of norepinephrine-equivalent to maintain systolic blood pressure > 90 mm Hg.
6. Impaired consciousness with a Glasgow coma score ≤ 12.
7. Patients with urgent need for intubation, including respiratory or cardiac arrest, respiratory pauses with loss of consciousness or gasping for air, severe hypoxemia defined as SpO2 lower than 90% despite maximal oxygen support.
8. Patients with contraindication to NIV according to the French consensus conference, patient refusal, cardiorespiratory arrest, coma, non-drained pneumothorax, unresolved vomiting, upper airway obstruction, hematemesis or severe facial trauma, thoracic or abdominal surgery in the previous 7 days.
9. A do-not-intubate order at time of inclusion.
10. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Intubation-free survival rate | From randomization to 28 days
  The proportion of patients who intubation-free and alive within 28 days after randomization.

SECONDARY OUTCOMES:
28-day mortality | From randomization to 28 days
  The proportion of patients who are died within 28 days
Intubation rate within 28 days | From randomization to 28 days
  The proportion of patients who are intubated within 28 days after randomization
A ranked composite score incorporating death and intubation through day 28 | From randomization to 28 days
  Priority sequence: 28-day mortality, followed by 28-day intubation
Meeting the prespecified criteria for intubation within 28 days. | From randomization to 28 days
  The proportion of patients who meeting the prespecified criteria for intubation within 28 days.
ICU mortality | From randomization to ICU discharge, assessed up to 60 days
  The proportion of patients who died within the ICU
In-hospital mortality | From randomization to hospital discharge, assessed up to 60 days
  The proportion of patients who died within the hospital
Change in Discomfort scale after 1 hour of randomization | Time from randomization to 1hour
  The discomfort scale are calculated using 100-mm visual-analogue scale
Invasive ventilator-free days at 28 days | From randomization to 28 days
  Days alive without endotracheal intubation and invasive mechanical ventilation
Circulatory support-free days at day 28 | From randomization to 28 days
  Circulatory support defined as infusion of any vasopressor/inotrope agent for a minimum of 1 hour (i.e. norepinephrine, epinephrine, phenylephrine, vasopressin analogues, angiotensin, dopamine, dobutamine, milrinone or levosimendan)
Time from randomization to an improvement of two points on a seven-category ordinal scale | From randomization to 28 days
  1, not hospitalized with resumption of normal activities; 2, not hospitalized, but unable to resume normal activities; 3, hospitalized, not requiring supplemental oxygen; 4, hospitalized, requiring supplemental oxygen; 5, hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both; 6, hospitalized, requiring ECMO, invasive mechanical ventilation, or both; and 7, death
ICU-free days at day 28 | From randomization to 28 days
  The number of ICU-free days within 28 days after randomization
Hospital-free days at day 28 | From randomization to 28 days
  The number of Hospital-free days within 28 days after randomization

OTHER OUTCOMES:
Vomiting | From randomization to 28 days
  The proportion of patients with vomiting, judged by the clinicians according to the clinical manifestations.
Aspiration of gastric contents | From randomization to 28 days
  The proportion of patients with aspiration of gastric contents, judged by the clinicians according to the clinical manifestations.
Nasal/facial skin necrosis | From randomization to 28 days
  The proportion of patients with nasal/facial skin necrosis, judged by the clinicians according to the clinical manifestations.
Pneumothorax | From randomization to 28 days
  Pneumothorax detected through chest X-ray or CT scan
Cardiac arrest | From randomization to 28 days
  The proportion of patients with cardiac arrest
Other adverse events | From randomization to 28 days
  The proportion of other adverse events related to the interventions assessed by investigators

CONTACTS AND LOCATIONS:
Overall Officials: Ling Liu, PhD, Study Director — Zhongda Hospital, School of Medicine, Southeast University
Locations (1):
- Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No